CLINICAL TRIAL: NCT06088238
Title: Use of Supramolecular Solvents in the Identification and Quantification of Substances of Very High Concern and Endocrine Disruptors Released From Michigan-type Occlusal Splints in Saliva: in Vitro and in Vivo Pilot Study.
Brief Title: Endocrine Disruptors in Saliva Released From Bruxism Splints.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidad Europea de Madrid (Other)
Collaborators: Universidad de Córdoba (Other); Universidade da Coruña (Other)
Responsible Party: Principal Investigator, Susana David Fernández, PhD, Universidad Europea de Madrid
Other Study IDs: 23.282
Record Dates: First submitted 2023-06-23; First posted 2023-10-18 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-06

CONDITIONS: Bruxism
Keywords: dental material; endocrine disruptor; substances of very high concern; saliva; occlusal splint; acrylic dental material
MeSH Terms: conditions — Bruxism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — SALIVA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The effects of endocrine disruptors (EDs) are well known. Therefore, the aim of this observational study is to analyse saliva samples from volunteers who request a bruxism splint, before, during and after fitting, to find out whether they are assimilated by the body, answering the following questions:

* Do Michigan-type splints release endocrine disruptors or substances of particular concern?
* In what concentration are they present in saliva?

Participants will be asked to take saliva samples at different times over a period of 6 months. This will also be accompanied by the relevant clinical and oral history. A previous in vitro study is required, which is complemented by an in vivo study. The methodology is new in dentistry: super solvents which, combined with liquid chromatography coupled to a mass spectrometer (LC-HRMS), allows a wider range of substances to be detected, in a more ecological and simpler way, as they are not organic solvents derived from petroleum. The splint is chosen because it is an everyday treatment, which is increasingly in demand, especially after the pandemic. It is subdivided into two types, depending on the method of manufacture: injected and printed (more ecofriendly).

DETAILED DESCRIPTION:
DESCRIPTION:

This is a prospective analytical observational analytical experimental pilot study with the aim of analysing substances of particular concern and endocrine disruptors detected in saliva, released by conventional dental devices, before and after the intervention. They will therefore be paired samples, where the control group will be the same subject, minimising the independent variables: saliva pH, microbiome, salivary flow, habits, occlusal wear, erosion by external agents and saliva.

Saliva sampling will be carried out according to the conventional protocol RD 1716/2011. The saliva containers will comply with the requirements of ISO 6717:2021. They shall be packaged and transported according to the protocol Order JUS/1291/2010 of 13 May. All samples shall be identified with the number assigned to the volunteer, time, material and type of manufacture (processed, machined or printed), and shall be sent to the Chemical Institute for Energy and Environment (IQUEMA). University of Cordoba, where they will be analysed by the SAC group, for subsequent statistical treatment and interpretation.

POPULATION AND SAMPLE CALCULATION. The sample will be obtained from patients who are registered in the database of the Polyclinic of the European University of Madrid, who request a Michigan type splint for the treatment of bruxism, made of acrylic, made in two of the usual ways: printed or injected, in accordance with the inclusion and exclusion criteria shown in Appendix I. As the samples are treated with an innovative methodology in the field of dentistry, such as super solvents, this is a pilot study in which two groups of 15 participants each are formed, depending on the manufacturing process of the splint: injected or printed, totalling 30 volunteers.

STUDY PERIOD Recruitment is expected to be completed in January 2024, and sample collection is expected to be completed in September 2024.

VOLUNTEER RECRUITMENT:

The study groups will be constituted according to the requirements and inclusion criteria. Each of the subjects will be informed of the purpose and methodology of the project by means of a volunteer information document (Annex II) and must sign the informed consent form provided for this purpose (Annex III); they may resign at any time to participate in the project. The data of the members will be stored in a medical record with an individual key number, in accordance with the regulations contained in the current Organic Law 3/2018, of 5 December, on the Protection of Personal Data.

Appointments will be made as follows:

APPOINTMENT 1: A conventional computerised clinical history is taken of the patient, in which data is collected on general health, orofacial, nutritional and hygiene habits. We explain in detail what the treatment consists of: Michigan type relaxation splint (device to prevent tooth wear due to bruxism). Each intervention is governed by scientific and deontological criteria, respecting all the ethical rules of research. The following is a detailed description of the study, its duration and methodology. The four moments of saliva collection will be explained: before, during, and 3 and 6 months after placement, as follows:

* Moment 0: the day of the appointment, before the intervention.
* Time 1: the day of the appointment, device placement.
* Time point 2: 3 months after device placement.
* Time 3: 6 months after treatment.

Information and informed consent will be given.

Appointment 2: Preparation and taking of models for the Michigan type splint according to the conventional protocol for this treatment.

APPOINTMENT 3: The models will be assembled in the articulator to send and request the making of the splint, specifying whether it is injected or printed.

APPOINTMENT 4: A saliva sample will be taken in the device for this purpose. The appliance will be fitted and occlusal adjustments will be made with a handpiece and conventional acrylic and polishing burs, after checking for proper fit and retention. After completion of the procedure, a new saliva sample shall be taken. The samples shall be identified with the patient's assigned code and stored according to conventional standards. An appointment will be made after 6 months to continue with the study and in accordance with the review times for proper oral health.

APPOINTMENT 5: The intraoral check-up will be carried out, checking the intraoral health and the state of the splint, with the pertinent adjustments, according to conventional protocol. A new saliva sample will be taken. The patient will be seen after 3 months.

APPOINTMENT 6: The intraoral check-up will be carried out, checking the intraoral health and the state of the splint, with the pertinent adjustments, according to conventional protocol. A new saliva sample will be taken. The period of sample collection for this subject will end.

Previously, the substances released by the specific material used to make the devices will be identified in the laboratory. The reason for this is the highly dynamic nature of the dental materials market. For this purpose, the solutions will be analysed by liquid chromatography coupled to a mass spectrometer (LC-HRMS). The identification of the compounds present will be based on a non-directed suspect screening approach, comparing the results obtained in the analyses with those already existing for the compounds included in the suspect list. This list will be compiled on the basis of the information gathered during the literature review, among other sources. Thus, it will range from compounds whose presence is expected such as those indicated by the manufacturer, to emerging compounds that might be present due to storage conditions, use, etc. For the identification, statistical and chemometric techniques will be used to establish the correlation between the analytical signals obtained in the LC-HRMS and the information (e.g. masses, structure, mass spectra, etc.) available in bibliography and publicly available spectrophotometric libraries (e.g. Mass Bank). In a second phase, the compounds identified in the first stage will be prioritised according to their level of identification, frequency of detection, toxicity (if known) and availability of analytical standards. Finally, quantification of these compounds will be carried out.

Thus, knowing the possible elements identified, the saliva samples can be treated. This is carried out with a volatile supramolecular solvent spontaneously synthesised by the addition of hexanol and tetrahydrofuran. The methodology to be followed is the same as previously described in the in vitro phase.

Dependent variables: substances of particular concern and endocrine disruptors. Independent variables: usual residence, type of manufacture (printed or injected), time, age, type of polymerisation.

After identification and quantification of the detected substances, the data will be collected in a database with the volunteer's information (ANNEX IV).

Finally, the results will be analysed and correlated with those obtained in the experimental laboratory phase, and the possible participating variables: age, type of manufacture and habits of the participant.

ELIGIBILITY:
Inclusion Criteria:

* To be of legal age
* Be able to attend Polyclinic for 6 months.
* Require an acrylic relaxation splint type Michigan
* Not be pregnant
* Not be breastfeeding

Exclusion Criteria:

* Be a minor
* Allergy to any type of plastic material, acrylic or resins for dental use.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — Female Male Other
Study Population: The sample will be obtained from patients who are registered in the database of the Polyclinic of the European University of Madrid, who request a Michigan type splint for the treatment of bruxism, made of acrylic, made in two of the usual ways: printed or injected, in accordance with the inclusion and exclusion criteria. As the samples were treated with an innovative methodology in the field of dentistry, such as super solvents, this is a pilot study in which two groups of 15 participants each were formed, depending on the manufacturing process of the splint: injected or printed, totalling 30 volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2024-09-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Identification of endocrine disruptors (EDs) or substances of concern of very high concern (SVHC)in saliva released by Michigan type occlusal splints before, during and after their application. | 6 months
  Treatment of samples by addition of hexanol and tetrahydrofuran. The solutions will be analysed by liquid chromatography coupled to a LC-HRMS mass spectrometer.
Quantification of endocrine disruptors or substances of very high concern (SVHC) in saliva released from Michigan type occlusal splints before, during and after application. | 6 months
  LC-HRMS (Liquid chromatography-high resolution mass spectrometry). Maximum dose recommended by the FDA (Food and Drug Administration): 4 micrograms/kilo/day in adults.

SECONDARY OUTCOMES:
Identification of endocrine disruptors or substances of very high concern (SVHC) released from Michigan-type occlusal splints in vitro simulating oral environment and wear. | 1 month
  Treatment of samples by addition of hexanol and tetrahydrofuran. The solutions will be analysed by liquid chromatography coupled to a LC-HRMS mass spectrometer
Quantification of endocrine disruptors (EDs) or substances of very high concern (SVHCs) released from Michigan-type occlusal splints simulating oral environment and wear and tear | 1 month
  LC-HRMS (Liquid chromatography-high resolution mass spectrometry). Maximum dose recommended by the FDA (Food and Drug Administration): 4 micrograms/kilo/day in adults.

OTHER OUTCOMES:
Relationship between concentrations of endocrine disruptors or substances of very high concern detected in vitro and in vivo | 1 month
  LC-HRMS (Liquid chromatography-high resolution mass spectrometry). Maximum dose recommended by the FDA (Food and Drug Administration): 4 micrograms/kilo/day in adults.
Differences in concentrations of endocrine disruptors or substances of very high concern released from injected and in vivo imprinted Michigan-type splints | 1 month
  LC-HRMS (liquid chromatography-high resolution mass spectrometry). Maximum dose recommended by the FDA (Food and Drug Administration): 4 micrograms/kilo/day in adults.

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT06088238/Prot_ICF_000.pdf